CLINICAL TRIAL: NCT06484569
Title: Effectiveness of Exercises Given Along With Ergonomics Training in Textile Workers: A Randomized Controlled Trial
Brief Title: Effectiveness of Exercises Given Along With Ergonomics Training in Textile Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar12
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Work Injury; Work-related Illness
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): They will receive ergonomics training
  Interventions: Other: Control
- exercise (Experimental): Ergonomics training, exercise training and cranio sacral therapy will be applied
  Interventions: Other: Control; Other: exercise and cranio sacral therapy

INTERVENTIONS:
Other: Control — The content of ergonomics training will include the definition of ergonomics, ergonomic positions and arrangements. Postural arrangements will be explained to patients individually and supported by a brochure.
Other: exercise and cranio sacral therapy — Posture exercises Stretching exercises Strengthening Exercises In addition, deep tissue massage will be applied to increase blood circulation and cranio-sacral therapy will be applied to increase cerebrospinal fluid circulation.
  Arms: exercise

SUMMARY:
The aim of this study is to investigate the effectiveness of ergonomic training and exercise training given to workers in a textile factory.

DETAILED DESCRIPTION:
The study will include workers between the ages of 18-60 who have neck pain and work at Ölmezler Textile Industry Trade limited company in Van province. Participants will be divided into two groups as experimental and control groups. All participants will receive ergonomic training. In addition, exercise training will be given to individuals in the experimental group. Exercises will be explained individually and will be supported with an exercise brochure. Craniosacral therapy will also be applied to the experimental group and a brochure will be given to teach joint protection principles. Participants will be asked to do the given exercises 3 days a week and continue for 12 weeks. The given exercises will be followed with an exercise follow-up chart. An evaluation will be made before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-60 years old
* Working full time
* Experiencing neck pain

Exclusion Criteria:

* Being under 18 or over 60 years old
* Presence of diseases accompanying neck pain
* Exercise intolerance
* Working part time

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Bournemouth Neck Pain Survey | 14 weeks
  The survey consists of 7 questions. In addition to questions about pain and disability, it also includes questions about psychosocial issues. Each question is scored between 0 and 10. The highest score is 70, with a higher score indicating a higher level of disability. The content of the survey consists of variables that must be questioned for individuals with neck pain, such as pain severity, the effect of pain on daily life activities and social life, anxiety-depression level, kinesiophobia and coping with pain.
The Fremantle Neck Awareness Questionnaire | 14 weeks
  The questionnaire is a Likert-type questionnaire (0 = Never/Never feel like this, 1 = Rarely feel like this, 2 = Sometimes or sometimes feel like this, 3 = Often feel like this, 4 = Always or most of the time feel like this) that evaluates individual-specific altered perception. The questionnaire asks individuals 9 questions such as how they perceive their neck in relation to their body, how they perceive their body position. The total score varies between 0-36. A high score indicates a poor prognosis.
Fatigue Severity Scale | 14 weeks
  The person indicates how much he or she agrees with each item by choosing numbers from 1 to 7. 1 means completely disagree, 7 means completely agree. The score range of the scale, which consists of 9 questions in total, is 9-63. A score of 36 or higher indicates severe fatigue.
Pittsburgh Sleep Quality Survey | 14 weeks
  The scale includes a total of 24 questions. 19 of these questions are self-evaluation questions, and 5 of them are answered by the individual's spouse or a roommate. These 5 questions are used for clinical information only and are not included in the scoring. The scale questions that determine sleep quality include various factors related to sleep quality. These questions are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems; 18 items were grouped as 7 component scores. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. The scale does not indicate the presence of sleep disorders or the prevalence of sleep disorders. However, it is stated that a total score of 5 and above indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal ATASOY, Study Chair — Uskudar University
Locations (1):
- Ölmezler Textile LTD.CO., Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Islam T. Health Concerns of Textile Workers and Associated Community. Inquiry. 2022 Jan-Dec;59:469580221088626. doi: 10.1177/00469580221088626. PMID 35604168
- [Background] Michaud F, Pazos R, Lugris U, Cuadrado J. The Use of Wearable Inertial Sensors and Workplace-Based Exercises to Reduce Lateral Epicondylitis in the Workstation of a Textile Logistics Center. Sensors (Basel). 2023 May 27;23(11):5116. doi: 10.3390/s23115116. PMID 37299843
- [Background] Metgud DC, Khatri S, Mokashi MG, Saha PN. An ergonomic study of women workers in a woolen textile factory for identification of health-related problems. Indian J Occup Environ Med. 2008 Apr;12(1):14-9. doi: 10.4103/0019-5278.40810. PMID 20040992
- [Background] Eraslan U, Gelecek N, Genc A. Effect of scapular muscle endurance on chronic shoulder pain in textile workers. J Back Musculoskelet Rehabil. 2013;26(1):25-31. doi: 10.3233/BMR-2012-0346. PMID 23411645
- [Background] Split W, Kotwica S, Woszczak M. [Role of exercise therapy in the prevention of lumbosacral backache in textile industry workers]. Med Pr. 1984;35(6):465-9. Polish. PMID 6242064
- [Derived] Atasoy H, Sevgin O, Karamancioglu B, Dikmen Hosbas B. Ergonomics training with exercise and manual therapy in textile workers: a randomized controlled trial. Int Arch Occup Environ Health. 2025 Sep;98(7):661-672. doi: 10.1007/s00420-025-02160-9. Epub 2025 Aug 14. PMID 40810742